CLINICAL TRIAL: NCT05634876
Title: A Phase 1b Clinical Trial of UB-312 in Patients With Synucleinopathies
Brief Title: UB-312 in Patients With Synucleinopathies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-00631
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple System Atrophy; Parkinson Disease
MeSH Terms: conditions — Multiple System Atrophy; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment First - MSA (Experimental): Includes participants with MSA only.
  Patients in the treatment-first arm will receive active treatment at weeks 1, 5, 13, 25, 37, 49, 73, and 97; and placebo doses at weeks 17, 61, 85, and 109. Participants will be followed up for 24 weeks after their last dose.
  All participants will receive three priming doses of UB-312 300 µg, followed by 5 booster doses of UB-312 300 µg. To keep the blind, both treatment arms will receive active treatment and placebo injections for a total of 12 injections (8 active treatment injections + 4 placebo injections).
  Interventions: Biological: UB-312 Injection; Biological: Placebo Injection
- Delayed Start - MSA (Experimental): Includes participants with MSA only
  Patients in the delayed-start arm will receive placebo injections at weeks 1, 5, 73, and 97; and active treatment at weeks 13, 17, 25, 37, 49, 61, 85, and 109. Participants will be followed up for 24 weeks after their last dose.
  All participants will receive three priming doses of UB-312 300 µg, followed by 5 booster doses of UB-312 300 µg. To keep the blind, both treatment arms will receive active treatment and placebo injections for a total of 12 injections (8 active treatment injections + 4 placebo injections).
  Interventions: Biological: UB-312 Injection; Biological: Placebo Injection
- Treatment First - PD (Experimental): Includes participants with PD only.
  Patients in the treatment-first arm will receive active treatment at weeks 1, 5, 13, 25, 37, 49, 73, and 97; and placebo doses at weeks 17, 61, 85, and 109. Participants will be followed up for 24 weeks after their last dose.
  All participants will receive three priming doses of UB-312 300 µg, followed by 5 booster doses of UB-312 300 µg. To keep the blind, both treatment arms will receive active treatment and placebo injections for a total of 12 injections (8 active treatment injections + 4 placebo injections).
  Interventions: Biological: UB-312 Injection; Biological: Placebo Injection
- Delayed Start - PD (Experimental): Includes participants with PD only.
  Patients in the delayed-start arm will receive placebo injections at weeks 1, 5, 73, and 97; and active treatment at weeks 13, 17, 25, 37, 49, 61, 85, and 109. Participants will be followed up for 24 weeks after their last dose.
  All participants will receive three priming doses of UB-312 300 µg, followed by 5 booster doses of UB-312 300 µg. To keep the blind, both treatment arms will receive active treatment and placebo injections for a total of 12 injections (8 active treatment injections + 4 placebo injections).
  Interventions: Biological: UB-312 Injection; Biological: Placebo Injection

INTERVENTIONS:
Biological: UB-312 Injection — UB-312, provided by Vaxxinity, contains 300 μg of p4573kb Drug Substance (synthetic peptide immunogen) formulated with CpG1 and Adju-Phos as a white, opaque, liquid suspension. The biological will be injected intramuscularly. The injection site will be the deltoid muscle.
Biological: Placebo Injection — Placebo will be injected intramuscularly. The injection site will be the deltoid muscle.

SUMMARY:
This is a Phase 1b study to determine the safety, tolerability, and immunogenicity of UB-312 in participants with multiple system atrophy (MSA), and in participants with Parkinson's disease (PD). UB-312 is a UBITh®-enhanced synthetic peptide-based vaccine and may provide an active immunotherapy option for treating synucleinopathies including the most prevalent form, PD; and the most rapidly progressive form, MSA.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is signed and dated by the participant.
2. Male or female aged 40 to 75 years old, inclusive, at screening.
3. Participants must have a body mass index (BMI) between 18 and 32 kg/m2, inclusive at screening, and with a minimum weight of 50 kg.
4. Expected to be able to undergo all study procedures.
5. Women must be of non-childbearing potential (postmenopausal for at least 12 months before screening or surgically sterile) or, if of childbearing potential, must be using medically acceptable contraceptive measures throughout the study and for at least 24 weeks after their last dose of study treatment.
6. Male participants and their partners of childbearing potential must commit to using medically acceptable contraception for the study duration and at least 90 days after their last dose of study treatment. Men must refrain from donating sperm during this same period. The female partners should use a medically acceptable contraception method, and these contraceptive measures should be used throughout the study and for at least 90 days after their last dose of study treatment.
7. A diagnosis of PD or MSA, confirmed by the PI, as per the current Movement Disorders Society's criteria (Postuma 2015, Wenning 2022).
8. Stable treatment of permitted antiparkinsonian medications from 30 days before first study drug administration or 60 days for MAO-B inhibitors and expected to remain stable throughout the study unless required adjustment or initiation per the investigator's judgment; except for short-acting rescue medications, which are allowed (see Section 7.1 for the list of permitted medications).
9. Eligible participants must be fully vaccinated against COVID-19 according to local guidelines. Participants also must have received a COVID-19 booster vaccination, and the interval between booster vaccination and sample collection for inflammatory markers at Screening should be at least seven days.
10. Subjects with a MOCA score > 21 at screening and throughout enrollment.

Exclusion Criteria:

1. Clinically significant abnormalities, as judged by the investigator, in test results (including hepatic and renal panels, complete blood count, chemistry panel, a level of anti-cyclic citrullinated peptide (anti-CCP) above the upper limit of normal (ULN) at Screening, positive antinuclear antibodies (ANA), except judged to be clinically irrelevant by the investigator, urinalysis, ECG and imaging), or vital signs. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant.
2. History of medical, neurological, or psychiatric conditions, which in the opinion of the investigator, may compromise the participant's safety or scientific value of the study, posing an unacceptable risk to the participant or interfering with the participant's ability to comply with the study procedures or abide by study restrictions.
3. History of Substance Use Disorder within the past 2 years before screening (Diagnostic and Statistical Manual of Mental Disorders-5 [DSM-V] criteria).
4. Acute or chronic infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) at Screening or any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV-1, HIV-2 infection, or cytotoxic therapy in the previous 5 years.
5. History or evidence of an autoimmune disorder (e.g. Sjogren's syndrome, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, etc.), which in the opinion of the investigator may compromise the patient's safety or scientific value of the study, posing an unacceptable risk to the participant.
6. History of anergy.
7. Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug or vaccine, or multiple drug allergies (non-active hay fever is acceptable).
8. History of cancer (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved) which has not been in remission for at least 5 years before Screening.
9. Contraindications to MRI, including but not limited to the presence of metal devices or implants (e.g., pacemaker, vascular- or heart-valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes.
10. Receipt of an investigational product or device, or participation in a drug research study within 90 days before baseline at V1.
11. Participated/participating in any clinical trial with monoclonal antibodies or vaccines directed at aSyn.
12. Underwent any procedures/studies involving intracranial surgery, implantation of a device into the brain, or stem cell study.
13. Pregnancy, confirmed by a positive pregnancy test.
14. Participants who are currently breastfeeding or intend to breastfeed during the study. Participants should not be willing to get pregnant and breastfeed till 24 weeks after the last injection.
15. Use of any prohibited medications within 30 days or 5 half-lives (whichever is greater) before Screening till the end-of-study; also excluded administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of Screening (including prednisone or equivalent, greater than or equal to 0.5 mg/kg/day; except Intranasal, inhalation, and topical steroids are allowed).
16. Immunization or vaccination will be prohibited within 2 weeks before Screening. Regular vaccinations scheduled for preventative illnesses (e.g., flu, COVID-19) required as per local guidelines after Screening until Week 16 need to be discussed with the Investigator and approved on a case-by-case basis. Vaccinations after Week 16 until the end of the study are allowed if not within 2 weeks of (e.g., 2 weeks before and 2 weeks after) each post-baseline IP administration.
17. Any contraindication to undergoing a lumbar puncture (e.g., anatomical variations or local skin infection), as judged by the investigator.
18. Loss or donation of blood over 500 mL within three months before Screening or intention to donate blood or blood products for transfusion during the study and 13 months after their last dose.
19. Received blood and/or blood derivatives treatment within 3 months before Screening.
20. Positive test result for SARS-CoV-2 infection (if test performed according to local guidelines) in the 2 weeks before the first dose.
21. Other known or suspected causes of Parkinsonism other than idiopathic PD or MSA, including but not limited to, progressive supranuclear gaze palsy, drug- or toxin-induced parkinsonism, essential tremor, primary dystonia, or vascular parkinsonism.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Serum Levels of anti-aSyn Antibodies from First Injection | Day 1, Week 133
  Derived from participant serum samples and calculated using a validated enzyme immunoassay.
Change in CSF Levels of anti-aSyn Antibodies from First Injection | Day 1, Week 133
  Derived from participant cerebrospinal fluid (CSF) samples and calculated using a validated enzyme immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Horacio.kaufmann@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Horacio.kaufmann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.